CLINICAL TRIAL: NCT06823635
Title: An International Multicenter Study on Transcatheter Device Closure of Perimembranous Ventricular Septal Defects
Acronym: PERI-CLOSE
Status: Not yet recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PERI-CLOSE
Record Dates: First submitted 2025-01-31; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Perimembranous Ventricular Septal Defect
Keywords: Cardiovascular Abnormalities; Congenital Heart Disease; Device Closure; Heart Defects, Congenital; Heart Septal Defects; Heart Septal Defects, Ventricular; Transcatheter Interventions; Ventricular Septal Defects
MeSH Terms: conditions — Cardiovascular Abnormalities; Heart Defects, Congenital; Heart Septal Defects; Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with perimembranous ventricular septal defects (PmVSDs) who provided informed consent and u
  Interventions: Device: Transcatheter device closure of perimembranous ventricular septal defects (PmVSDs)

INTERVENTIONS:
Device: Transcatheter device closure of perimembranous ventricular septal defects (PmVSDs) — Transcatheter closure of perimembranous ventricular septal defects (PmVSDs) using an occluder device either specifically designed for this purpose or used off-label.

SUMMARY:
The international multicenter registry aims to gather real-world data on patient outcomes and assess the procedural success and performance of various device occluders used in the transcatheter treatment of pediatric and adult patients with perimembranous ventricular septal defects (PmVSD).

DETAILED DESCRIPTION:
This is a non-randomized, multicenter, international, non-interventional, observational, retrospective post-marketing clinical follow-up study designed to evaluate the feasibility, safety, and efficacy of transcatheter closure of perimembranous ventricular septal defects (PmVSD) using commercially available device occluders, whether specifically designed for this purpose or used off-label.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with perimembranous ventricular septal defects (PmVSD), as defined by 2D transthoracic echocardiography according to previously published classifications.
2. Defect size between 3 mm and <20 mm on the left ventricular side, as measured by 2D echocardiography.
3. Left-to-right ventricular shunt.
4. Age ≥3 months and body weight≥5 kg.
5. Symptomatic patients (heart failure, failure to thrive, recurrent respiratory infections, and rest or exercise dyspnea) or asymptomatic patients with progressive heart enlargement.
6. History of infective endocarditis related to the PmVSD or hemodynamically significant PmVSD with: Qp/Qs >1.5 on catheterization, left ventricular volume overload (LVEDD z-score >2) based on echocardiography, or pulmonary hypertension on catheterization (mean pulmonary artery pressure >20 mmHg).
7. Presence or absence of aortic valve prolapse, with or without regurgitation.
8. Presence or absence of a membranous septal aneurysm, with or without inlet or outlet extension.

Exclusion Criteria:

1. Eisenmenger physiology (pulmonary vascular resistance > 8 Wood units, nonreactive) with an exclusive right-to-left shunt.
2. Pre-existing complete heart block or high-risk proximity of the conduction system to the defect without prior pacemaker implantation.
3. Severe aortic or tricuspid valve disease requiring surgical or catheter-based intervention.
4. Pregnancy or planned pregnancy if the procedure involves X-ray exposure.
5. Extensive congenital cardiac anomalies requiring surgery.
6. Thrombus at the implant site or documented venous thrombus in access vessels.
7. Sepsis, active endocarditis, or bacterial infections within one month pre-procedure.
8. Uncontrolled bleeding or clotting disorders.
9. Contraindications to antiplatelet therapy or refusal of blood transfusions.
10. Cardiac malformations dependent on the presence of a perimembranous ventricular septal defect (PmVSD).
11. Lack of informed written consent for the procedure
12. Failure to attend any follow-up visit post-discharge.
13. Patients under guardianship or curatorship
14. Patients deprived of liberty
15. Patients under court protection
16. Patients or legal guardians refusing the use of personal data for this research

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients, regardless of gender or geographical location, with perimembranous ventricular septal defects (PmVSDs) who provided informed consent and underwent transcatheter closure using commercially available occluder devices, whether specifically designed for this purpose or used off-label, were followed according to local hospital protocols.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Twelve-month composite non-hierarchical clinical success | From implant attempt to 12 hours post-procedure
  Defined as meeting the following 3 criteria: 1) technical success (device successfully implanted and retained at hospital discharge), 2) closure success (trivial or no residual shunt through 12 months), 3) safety success (no serious adverse events (SAEs) through 30 days, and no device events (removal or reintervention) through 12 months).
Technical success | From implant attempt to 12 hours post-procedure
  Successful device deployment and stable device position confirmed via post-procedure transthoracic echocardiography (TTE).
Closure success | From implant attempt to 12 hours post-procedure
  Complete shunt occlusion or trivial shunt on post-procedure TTE
Procedural success | From implant attempt to 12 hours post-procedure
  Technical success with complete closure of PmVSD (residual shunt ≤2 mm confirmed on post-procedure TTE), no interference with adjacent structures, including aortic and tricuspid valves.
Clinical success | From implant attempt to 12-month post-procedure
  In symptomatic patients: Resolution of patient-reported clinical symptoms (reduced fatigue, improved exercise tolerance) within 30 days, along with normalization of left ventricular dimensions on cardiac ultrasound, and/or a ≥20% reduction in pulmonary artery pressure from baseline.
Freedom from procedure or device-related major adverse events | From implant attempt to 12-month post-procedure
  Absence of procedure or device-related major adverse events, including:
  * Device migration or embolization requiring catheter or surgical intervention.
  * Complete heart block requiring permanent pacemaker implantation, device removal, or other medical treatment.
  * Severe aortic or tricuspid regurgitation (≥ moderate grade) requiring device removal, close monitoring, or intervention.
  * Life-threatening bleeding or significant vascular injury requiring catheter or surgical intervention.
  * Thrombosis of device or vascular access that requires device removal, thrombolytic therapy, catheter, or surgical intervention.
  * Severe acute hemolysis, requiring blood transfusion device removal, catheter, or surgical intervention.

SECONDARY OUTCOMES:
Short-term complications (≤30 days) | From implant attempt to 30 days post-procedure
  Minor vascular complications (hematoma, pseudoaneurysm, minor bleeding). Transient arrhythmias (supraventricular tachycardia, non-sustained VT, first-degree AV block).
Long-term outcomes | From implant attempt to 60-month post-procedure
  * Sustained complete closure (no or minimal residual shunt on TTE).
  * Late-onset device-related complications (new-onset aortic or tricuspid regurgitation, delayed second-degree or complete heart block, or arrhythmias requiring permanent treatment).
  * Device migration or embolization requiring catheter or surgical removal
  * Thromboembolism: thrombosis of device or vascular access that requires thrombolytic therapy
  * Hemolysis requiring prolonged or redo hospitalization and severe acute hemolysis requiring blood transfusion with or without intervention.
  * Death
Rate of incomplete closure at the 24-month follow-up. | From implant attempt to 24-month post-procedure
  Rate of incomplete closure at the 24-month follow-up: A significant shunt will be defined as ≥ moderate or requiring treatment (surgical or interventional). The residual shunt will be assessed using color Doppler echocardiography, with shunt size categorized according to previously published classifications.
Functional and quality-of-life measures | From implant attempt to 48-month post-procedure
  Improvement in NYHA/ROSS functional class and in pediatric patients, catch-up growth.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond N. Haddad, MD, MHSc, Principal Investigator — Marie Lannelongue Hospital
Locations (18):
- Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark
- France (4):
  - University Hospital of Bordeaux, Bordeaux
  - Marie Lannelongue Hospital, Le Plessis-Robinson
  - Lille University Hospital, Lille
  - Toulouse University Hospital, Toulouse
- University Children's Hospital, Tübingen, Germany
- National Cardiovascular Center of Harapan Kita, Jakarta, Indonesia
- Rajaie Cardiovascular, Medical and Research Center, Tehran, Iran
- Hôtel-Dieu de France University Medical Center, Beirut, Lebanon
- Hospital de Especialidades Pediátricas, Chiapas, Mexico
- The Children's Hospital, Lahore, Pakistan
- Silesian Center for Heart Diseases, Zabrze, Poland
- Madinah Cardiac Center MCC, Madinah, Saudi Arabia
- Turkey (Türkiye) (4):
  - Ankara City Hospital, Ankara
  - Koç University, Istanbul
  - Umraniye Training and Education Hospital, Istanbul
  - SBU Tepecik Training and Research Hospital, Izmir
- Al Jalila Children's Speciality Hospital, Dubai, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No